CLINICAL TRIAL: NCT01756430
Title: A Randomized, Double-blind, Multi-center, Phase 3 Trial to Evaluate the Efficacy and Safety of Carvedilol SR Versus Carvedilol IR in Patients With Essential Hypertension
Brief Title: Efficacy and Safety of Carvedilol SR Versus Carvedilol IR in Patients With Essential Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 125HT12001
Record Dates: First submitted 2012-12-20; First posted 2012-12-27 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Hypertension
Keywords: Carvedilol SR; Carvedilol IR; Hypertension; Essential Hypertension
MeSH Terms: conditions — Hypertension; Essential Hypertension | interventions — Carvedilol; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carvedilol SR 32mg, 64mg (Experimental): •Carvedilol SR 32mg QD for first 4 weeks and Carvedilol SR 64mg QD for following 4 weeks.
  Interventions: Drug: Carvedilol SR 32mg, QD; Drug: Carvedilol SR 64mg, QD
- Carvedilol IR 25mg (Active Comparator): •Carvedilol IR 25mg QD for first 4 weeks and Carvedilol IR 25mg BID for following 4 weeks.
  Interventions: Drug: Carvedilol IR 25mg, QD; Drug: Carvedilol IR 25mg, BID

INTERVENTIONS:
Drug: Carvedilol SR 32mg, QD — * Carvedilol SR 32mg QD for 4 weeks
  * With the others investigation product placebo 1 capsule QD and 1 tablet BID for 4 weeks.
  Other Names: Dilatrend SR
  Arms: Carvedilol SR 32mg, 64mg
Drug: Carvedilol SR 64mg, QD — * Carvedilol SR 64mg QD for 4 weeks
  * With the others investigation product placebo 1 capsule QD and 1 tablet BID for 4 weeks.
  Other Names: Dilatrend SR
  Arms: Carvedilol SR 32mg, 64mg
Drug: Carvedilol IR 25mg, QD — * Carvedilol IR 25mg QD for 4 weeks
  * With the others investigation product placebo 2 capsules and 1 tablet QD for 4 weeks.
  Other Names: Dilatrend IR
  Arms: Carvedilol IR 25mg
Drug: Carvedilol IR 25mg, BID — * Carvedilol IR 25mg BID for 4 weeks
  * With the others investigation product placebo 2 capsules QD for 4 weeks.
  Other Names: Dilatrend IR
  Arms: Carvedilol IR 25mg

SUMMARY:
The aim of present study is to evaluate the efficacy and safety of Carvedilol SR versus Carvedilol IR in Patients With Essential Hypertension

DETAILED DESCRIPTION:
* In patients with Essential hypertension to evaluate the efficacy and safety of Carvedilol SR (32mg, 64mg) or Carvedilol IR (25mg QD, 25mg BID) during 8 weeks.
* This study is consist of placebo run-in period(2~4 weeks_single blind) and treatment period(8 weeks_double blind).

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* at the screening visit(visit 1)

  * antihypertensive drugs not taking: 90mmHg ≤ mean sitDBP ≤ 109mmHg and mean sitSBP < 180mmHg
  * antihypertensive drugs taking: mean sitDBP ≤ 104mmHg and mean sitSBP < 180mmHg
* at the randomization visit(visit 2): 90mmHg ≤ mean sitDBP ≤ 109mmHg and mean sitSBP < 180mmHg
* willing and able to provide written informed consent

Exclusion Criteria:

1. At Screening, difference in measured blood pressure of the selected arm(sitDBP ≥ 10mmHg or sitSBP ≥ 20mmHg)
2. known or suspected secondary hypertension(ex. aortic coarctation, Primary hyperaldosteronism, renal artery stenosis, pheochromocytoma)
3. Type I Diabetes Mellitus, Type II Diabetes Mellitus with poor glucose control as defined by fasting glucosylated hemoglobin(HbA1c > 9%)
4. Corresponding to the following

   * has severe heart disease(Heart failure NYHA functional class 3, 4)
   * ischaemic heart diseases within 6 months (unstable angina or myocardial infarction)
   * myocardiopathy
   * Cor pulmonale
   * aortic stenosis , aortic valvular stenosis , mitral stenosis
   * abnormality of the conduction system as 2nd degree AV block, Complete AV block, Sick Sinus Syndrome, Sinus Block(In particular, pulse <50beats / min)
   * has heart attack with complication.
5. has cerebrovascular disease as cerebral infarction, cerebral hemorrhage within 6 months
6. has edema glottitis, allergic rhinitis, Respiratory diseases as Asthma, Chronic Obstructive Pulmonary Disease.
7. Peripheral circulatory disturbance( ex. Raynaud syndrome, intermittent claudication)
8. Fluid retention or overload to required intravenous inotropes.
9. known severe or malignant retinopathy(retinal hemorrhage, visual disturbance, Retinal microaneurysms and so on within 6 months)
10. defined by the following laboratory parameters:

    * hepatic dysfunction(AST/ALT ≥ UNL X 3)
    * renal dysfunction(serum creatinine ≥ UNL X 2)
11. any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of investigational products(ex. gastrointestinal tract surgery such as gastrectomy, gastroenterostomy or bypass, active inflammatory bowel syndrome within 12 months prior to screening, gastric ulcers need to treatment, gastrointestinal/rectal bleeding, impaired pancreatic function such as pancreatitis, obstructions of the urinary tract or difficulty in voiding)
12. history of drug or alcohol dependency within 6 months
13. premenopausal women(last menstruation < 12 months) not using adequate contraception, pregnant or breast-feeding
14. chronic inflammatory status need to treatment
15. known hypersensitivity related to carvedilol
16. history of malignancy including leukemia and lymphoma within the past 5 years
17. administration of other study drugs within 28 days prior to the first IP administration
18. in investigator's judgment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2012-12; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Mean Sitting Diastolic Blood Pressure (MSDBP) | After 4 and 8 weeks of treatment

SECONDARY OUTCOMES:
Mean Sitting systolic Blood Pressure (MSSBP) | After 4 weeks and 8 weeks of treatment
Control Rate | After 8 weeks of treatment
  Sitting DBP<90mmHg, Sitting SBP<140mmHg
Response Rate | After 8 weeks of treatment
  Reduction of Sitting DBP≥10mmHg, Sitting SBP ≥20mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Soon Kill Kim, Principal Investigator — The Hanyang Universitiy Guri Hospital; Sang-Hyun Ihm, Principal Investigator — The Catholic University of Korea Bucheon St.Mary's Hospital; Sang Hong Haek, Principal Investigator — The Catholic University of Korea, Seoul St. Vincent's Hospital; Jin-Bae Kim, Principal Investigator — Kyunghee University Medical Center; Dong Woon Jeon, Principal Investigator — National Health Insurance Service Ilsan Hospital; Chang-Wook Nam, Principal Investigator — Keimyung University, Donsan Hospital; Dong-Ju Choi, Principal Investigator — Seoul National University Bundang Hospital; Min Su Hyon, Principal Investigator — Soon Chun Hyang University Hospital; Young Jin Choi, Principal Investigator — Sejong General Hospital; Hyuck Moon Kwon, Principal Investigator — Gangnam Severance Hospital; Geu Ru Hong, Principal Investigator — Severance Hospital; Byung-Su Yoo, Principal Investigator — Wonju Severance Christian Hospital; Ji-Hyun Lim, Principal Investigator — Jesus hospital; Young Keun Ahn, Principal Investigator — Chonnam National University Hospital; Jin Ho Shin, Principal Investigator — Hanyang University Seoul Hospital
Locations (1):
- The Hanyang Universitiy Guri Hospital, Guri-si, Gyeonggi-do, South Korea